CLINICAL TRIAL: NCT05874570
Title: Doxycycline-containing Bismuth Quadruple Therapy for Helicobacter Pylori Rescue Treatment: a Randomized Controlled Trial
Brief Title: Doxycycline for Helicobacter Pylori Rescue Treatment
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rjhy20230002
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; rescue therapy; doxycycline; tetracycline
MeSH Terms: interventions — Esomeprazole; Tetracycline; Doxycycline; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tetracycline Bismuth Quadruple Therapy (Active Comparator): Esomeprazole 20mg bid, Bismuth Potassium Citrate 110mg qid, Tetracycline 500mg qid, Metronidazole 400mg qid
  Interventions: Drug: Esomeprazole; Drug: Bismuth Potassium Citrate; Drug: Tetracycline; Drug: Metronidazole
- Doxycycline Bismuth Quadruple Therapy (Experimental): Esomeprazole 20mg bid, Bismuth Potassium Citrate 110mg qid, Doxycycline 100mg bid, Metronidazole 400mg qid
  Interventions: Drug: Esomeprazole; Drug: Bismuth Potassium Citrate; Drug: Doxycycline; Drug: Metronidazole

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
Drug: Tetracycline — Antibiotics for H. pylori eradication
  Arms: Tetracycline Bismuth Quadruple Therapy
Drug: Doxycycline — Antibiotics for H. pylori eradication
  Arms: Doxycycline Bismuth Quadruple Therapy
Drug: Metronidazole — Antibiotics for H. pylori eradication

SUMMARY:
Current guidelines have recommended classical bismuth-containing quadruple therapy including proton-pump inhibitor, bismuth, tetracycline, metronidazole as the empirical rescue therapy. However, tetracycline is clinically unavailable in China and the high frequency of adverse events of bismuth quadruple therapy often result in poor compliance, which limited the applicability of this recommendation. This study aimed to compare the efficacy and tolerability of a 14-day bismuth-containing quadruple rescue therapy in which tetracycline was replaced by doxycycline.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection and with previous treatment failure

Exclusion Criteria:

* subjects naive to H. pylori treatment,
* under 18 or over 80 years old
* history of gastrectomy
* pregnant or lactating women
* severe systemic diseases or malignancy
* administration of antibiotics, bismuth, antisecretory drugs, or Chinese herb medicine in the preceding 8 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities)
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No